CLINICAL TRIAL: NCT04400500
Title: Approaches to Differential Diagnosis and Risk Stratification in Patients Hospitalized With Suspected Acute Coronary Syndrome Without Persistent ST-segment Elevation
Brief Title: Differential Diagnosis and Risk Stratification in Patients With Suspected NSTEACS
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 01-02/20
Record Dates: First submitted 2020-04-23; First posted 2020-05-22 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
Keywords: Non ST segment Elevation Acute Coronary Syndrome; Diagnosis; Prognosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — hsTn, NT-proBNP, hsCPR, cardiac FABP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected NSTEACS: Patients urgently admitted to the CCU with suspected NSTEACS
  Interventions: Diagnostic Test: Approaches to differential diagnosis and risk stratification

INTERVENTIONS:
Diagnostic Test: Approaches to differential diagnosis and risk stratification — Detailed analysis of clinical course, ECG, biomarkers (hsTn I, CK-MB mass, myoglobin, NT-proBNP, hsCPR, cardiac FABP on admission and after 3 hours; hsTn I, CK-MB mass and myoglobin after 6 hours if needed) as well as HEART, ADAPT, EDACS, T-MACS, GRACE, ACTION and TIMI scores.

SUMMARY:
To evaluate possibilities of rapid differential diagnosis and risk stratification in patients urgently admitted to the CCU with a suspected acute coronary syndrome without persistent ST-segment elevation (NSTEACS).

DETAILED DESCRIPTION:
Single centre prospective non-randomised non-comparative study of patients delivered by ambulance and admitted to the CCU with suspected NSTEACS.

Aims of this study are:

1. To characterize the contingent of patients admitted to the CCU with suspected NSTEACS.
2. To evaluate possibilities of fast differential diagnosis and risk stratification in patients admitted to the CCU with suspected NSTEACS using clinical data, ECG, biomarker levels (hsTn, NT-proBNP, hsCPR, cardiac FABP) as well as HEART, ADAPT, EDACS, T-MACS, GRACE, ACTION and TIMI scores.
3. To evaluate the correlation between clinical data, ECG, biomarker levels (hsTn, NT-proBNP, hsCPR, cardiac FABP) as well as HEART, ADAPT, EDACS, T-MACS, GRACE, ACTION and TIMI scores with presence and severity of coronary atherosclerosis in patients admitted to the CCU (intensive care unit) with suspected NSTEACS.

ELIGIBILITY:
Inclusion Criteria:

1. Delivered by ambulance to the CCU with suspected diagnosis "acute coronary syndrome (ACS)".
2. Signed informed consent.

Exclusion Criteria:

1. ACS with persistent ST-segment elevation.
2. Moribund; extremely severe condition on admission with a potentially unfavourable prognosis (cardiogenic shock, coma, cardiac arrest, an urgent need for mechanical ventilation).
3. Overt non-cardiac cause of clinical manifestations at the time of admission (bleeding, pulmonary embolism, aortic dissection, stroke).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients delivered by ambulance and admitted to the CCU with suspected diagnosis "acute coronary syndrome (ACS)".
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes | 6 monts
  Composite of death, (re) infarction, stroke or re-hospitalization
Final diagnosis | Up to 1 monts
  Final diagnosis - the main reason for urgent hospitalization - according to hospital case history

SECONDARY OUTCOMES:
Death | 6 months.
  Death upon discharge and up to 6 months
(re) infarction | Up to 1 monts
  (re) infarction upon discharge and up to 6 months
Stroke | 6 months.
  Stroke upon discharge and up to 6 months
Re-hospitalization | 6 months.
  Recurrent hospital admissions after discharge form the index hospitalization

OTHER OUTCOMES:
Urgent revascularisation | Up to 1 monts
  Revascularisation performed due to sudden clinical deterioration
Other adverse events | 6 months.
  All adverse events/complications not included in clinical outcomes end points.

CONTACTS AND LOCATIONS:
Overall Officials: Igor S Yavelov, PhD, Principal Investigator — National Medical Research Center for Therapy and Preventive Medicine
Locations (1):
- Eramishantsev Hospital, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No